CLINICAL TRIAL: NCT02135835
Title: A Multicentre, Parallel-Group, Randomised, Double-Blind Study to Evaluate the Efficacy and Safety of Shenfu Zhusheye in Patients With Acute Heart Failure.
Brief Title: A Study to Evaluate the Efficacy and Safety of Shenfu Zhusheye in Patients With Acute Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China Resources Sanjiu Medical & Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1312-Z-SHFU-ZS-RE
Record Dates: First submitted 2014-04-22; First posted 2014-05-12 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-01

CONDITIONS: Acute Heart Failure
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Shenfu Zhusheye (Experimental): 80 ml Shenfu Zhusheye + 70 ml 5% glucose injection, ivdrip, once a day for 7 days.
  Interventions: Drug: Shenfu Zhusheye; Drug: 5% glucose injection
- 5% glucose injection (Placebo Comparator): 150 ml 5% glucose injection, ivdrip, once a day for 7 days.
  Interventions: Drug: 5% glucose injection

INTERVENTIONS:
Drug: Shenfu Zhusheye
  Arms: Shenfu Zhusheye
Drug: 5% glucose injection

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Shenfu Zhusheye in patients with acute heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Acute Heart Failure according to Guidelines for the diagnosis and treatment of acute heart failure 2010 of Chinese Medical Association(Participants whose Heart function grade of NYHA is Ⅲ～Ⅳ).
* LVEF≤40%.
* NT-pro-BNP ≥1400 pg/mL or BNP ≥ 350pg/mL.
* Ages 18-80, male or female.
* All participants signed the informed consent.

Exclusion Criteria:

* Participants with abnormal liver function (ALT, AST≥3 times of upper limit of normal) or abnormal kidney function( Cr≥1.5 times of upper limit of normal or Cr >3.0 mg/dl (> 265 µmol/L)).
* SBP ≥ 150mmHg.
* Participants with severe chronic asthmatic bronchitis or acute episode of lung diseases.
* Participants with acute coronary syndrome, cardiogenic shock, aortic dissection, pulmonary embolism, severe ventricular arrhythmias, complete atrioventricular block without cardiac pacemaker, hypertrophic obstructive cardiomyopathy, restrictive cardiomyopathy and severe valvular disease without surgery.
* Participants with advanced cancer.
* Breastfeeding, pregnant and potentially fertile women participant.
* Participants with insanity.
* Known allergies with Shenfu Zhusheye or its ingredients in the past.
* Participants who have taken part in other clinical trials in last month.
* Participants who abuse alcohol or other drugs in last year.
* Participants who are not suitable for clinical trial under doctors' consideration.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2014-09-03 (Actual); Primary Completion 2017-03-24 (Actual); Study Completion 2017-03-24 (Actual)

PRIMARY OUTCOMES:
Proportion of patients whose NT - proBNP level reduce more than 30% compared to pre-treatment. | 0, 7 days

SECONDARY OUTCOMES:
Decrease rate in NT-proBNP compared to pre-treatment. | 0, 7 days.
Decrease value in NT-proBNP compared to pre-treatment. | 0, 7 days.
Likert rating scale of Dyspnoea. | 0, 7 days.
The results of Transthoracic Doppler-echocardiography . | 0, 7 days.
  Left ventricular ejection fraction (LVEF) and Left Ventricular Diastolic End Diameter (LVDED) will be measured with Transthoracic Doppler-echocardiography.
Heart function grade of NYHA. | 0, 7 days.
Composite endpoints. | Composite endpoints will be assessed during medication period and 28 days after medication.
  Composite endpoints were defined as death, cardiac arrest with resuscitation, readmission for heart failure, worsening heart failure with an intravenous pharmacologic agent for more than 4 hours, stroke or cases where the patient ceased active treatments because of worsening heart failure.
Safety assessments will be based on adverse event reports and the results of clinical laboratory tests, electrocardiogram. | Adverse event reports will be assessed during medication period and 28 days after medication. Clinical laboratory tests will be assessed at 0, 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Jiefu Yang, Principal Investigator — Beijing Hospital
Locations (25):
- China (25):
  - An Hui Provincial Hospital, Hefei, Anhui
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Fourth People's Hospital of Shenzhen（Futian Hospital）, Shenzhen, Guangdong
  - Daqing peoples hospital, Daqing, Heilongjiang
  - Nanshi Hospital of Nanyang, Nanyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Fouth Affiliated Hospital of China Mdical University, Shenyang, Liaoning
  - The People's Hospital of Liao Ning Province, Shenyang, Liaoning
  - Tongren Hospital Shanghai Jiao Tong University School Of Medicine, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital Of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Hospital (T.C.M.) Affiliated to Sichuan Medical, Luzhou, Sichuan
  - The Second People's Hospital of Yibin, Yibin, Sichuan
  - The First Affiliated Hospital of the Medical College,Shihezi University, Shihezi, XIjiangweiwuerzizhiqu
  - The First Affiliated Hospital of Xinjiang Medical, Ürümqi, Xinjiang
  - The Second Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiangweiwuerzizhiqu
  - Tongde hospital of Zhejiang Province, Hangzhou, Zhejiang
  - Beijing Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - Shang Hai Chest Hospital Shanghai JiaoTong University, Shanghai